CLINICAL TRIAL: NCT05588011
Title: Influence of Oxygenator Selection on Platelet Function and Rotational Thromboelastometry Following Cardiopulmonary Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BRADEN DULONG (Other)
Responsible Party: Sponsor-Investigator, BRADEN DULONG, Anesthesiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NSH REB# 1027560
Record Dates: First submitted 2022-10-06; First posted 2022-10-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Platelet Dysfunction; Cardiopulmonary Bypass
Keywords: Rotem; Plateletworks; Cardiopulmonary Bypass; Platelets; Platelet function; Oxygenator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LivaNova Inspire (Active Comparator): A high pressure oxygenator (LivaNova) will be used during cardiopulmonary bypass.
  Interventions: Device: LivaNova
- Terumo (Active Comparator): A low pressure oxygenator (Terumo) will be used during cardiopulmonary bypass.
  Interventions: Device: Terumo

INTERVENTIONS:
Device: Terumo — A low pressure oxygenator (Terumo) will be used during cardiopulmonary bypass.
  Arms: Terumo
Device: LivaNova — A high pressure oxygenator (LivaNova) will be used during cardiopulmonary bypass.
  Arms: LivaNova Inspire

SUMMARY:
Open-heart surgery requires temporarily stopping the heart and lungs and diverting the patient's blood to an outside system that takes over the function of the heart and lungs. This is possible through the use of cardiopulmonary bypass (CPB) which diverts blood, through plastic tubing, to a heart-lung machine which includes an oxygenator. The external oxygenator works as an artificial lung. This allows cardiac surgeons to operate in a field that is free of blood, while the patient's body continues to receive healthy blood.

CPB is an advanced medical technology that allows for heart surgeries, such as coronary artery bypass, heart valve surgery, and procedures involving major blood vessels. It is recognized that there are many risks associated with its use, including microscopic stress exerted on blood components by the oxygenator and tubing, which can lead to irreversible damage to the blood cells. This effect can contribute to bleeding during and after surgery. This type of bleeding can be difficult to monitor and treat, especially given the limited access to point-of-care blood testing to inform clinicians on what part of the blood is failing to function properly.

The investigators will use a point-of-care machine called Plateletworks to test the function of platelets during surgeries which require CPB. Platelets are an important part of blood that help stop bleeding by forming clots. At the investigators' institution two oxygenators are currently used interchangeably. These oxygenators have different properties that may impact how platelets function. This project will help determine if using a higher pressure oxygenator increases the risk of patients bleeding. Additionally, the investigators will compare the platelet data from Plateletworks to data collected from rotational thromboelastometry (ROTEM). This will yield valuable data about commonly used oxygenators and tests which can ultimately improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for non emergent cardiac surgery
* Anticipated long CPB time (Multi-vessel CABG, multi-valve surgeries, or combined CABG and valve procedures)

Exclusion Criteria:

* Pregnancy
* Age under 18 years on the surgery date
* Weight less than 60kg
* Any known pre-existing bleeding disorder
* Inability to provide informed consent
* Pre-existing abnormal fibrinogen level (normal: 1.8-4.7g/l)
* Significant liver disease (alanine aminotransferase or aspartate aminotransferase > 150 U/l)
* INR > 1.4
* PTT greater than 38 (off IV heparin for 12h prior to testing)
* Direct oral anticoagulant (DOAC) use within 72h preoperatively
* Significant renal disease (eGFR < 50)
* Emergency surgery
* Intake of anti-platelet drugs (including ticagrelor and Plavix but excluding ASA) within three days (72h) preoperatively
* Anemia (Hb < 110)
* Deep vein thrombosis (DVT) (within 3 months prior to OR)
* Pulmonary embolism (within 3 months prior to OR)
* Stroke (within 3 months prior to OR)
* Planned hypothermia below 28 degrees Celsius.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Plateletworks change in functional platelets | 24 hours from start of surgery (measured at the start and the end of cardiopulmonary bypass)
  Change in functional platelets during cardiopulmonary bypass as measure by Plateletworks. ((Functional Platelets start - Functional Platelets end) / Functional Platelets start) *100%.
Plateletworks functional platelet count | 24 hours from start of surgery (measured at the end of cardiopulmonary bypass)
  Functional platelet count at the end of cardiopulmonary bypass as measured by Plateletworks.
Percentage of platelets which are functional at the end of cardiopulmonary bypass | 24 hours from start of surgery (measured at the end of cardiopulmonary bypass)
  Percentage of platelets which are functional at the end of cardiopulmonary bypass as measured by Plateletworks.

SECONDARY OUTCOMES:
ROTEM change in functional platelets | 24 hours from start of surgery (measured at the start and the end of cardiopulmonary bypass)
  ROTEM platelet function = EXTEM A10 - FIBTEM A10. ROTEM change in functional platelets = ((ROTEM Functional Platelets start - ROTEM Functional Platelets end) / ROTEM Functional Platelets start) *100%.

OTHER OUTCOMES:
Change in functional platelets per unit time on cardiopulmonary bypass | 24 hours from start of surgery (measured at the start and the end of cardiopulmonary bypass)
  Change in functional platelets per unit time on cardiopulmonary bypass for each oxygenator. As measured by Plateletworks. (Functional Platelets start - Functional Platelets end / time on cardiopulmonary bypass).

CONTACTS AND LOCATIONS:
Overall Officials: Braden Dulong, MD, Principal Investigator — Nova Scotia Health
Locations (1):
- Halifax Infirmary site, Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Background] Despotis G, Eby C, Lublin DM. A review of transfusion risks and optimal management of perioperative bleeding with cardiac surgery. Transfusion. 2008 Mar;48(1 Suppl):2S-30S. doi: 10.1111/j.1537-2995.2007.01573.x. No abstract available. PMID 18302579
- [Background] Hardwick RA, Hellums JD, Peterson DM, Moake JL, Olson JD. The effect of PGI2 and theophylline on the response of platelets subjected to shear stress. Blood. 1981 Oct;58(4):678-81. PMID 7023570
- [Background] Karkouti K, McCluskey SA, Callum J, Freedman J, Selby R, Timoumi T, Roy D, Rao V. Evaluation of a novel transfusion algorithm employing point-of-care coagulation assays in cardiac surgery: a retrospective cohort study with interrupted time-series analysis. Anesthesiology. 2015 Mar;122(3):560-70. doi: 10.1097/ALN.0000000000000556. PMID 25485470
- [Background] Karkouti K, Callum J, Wijeysundera DN, Rao V, Crowther M, Grocott HP, Pinto R, Scales DC; TACS Investigators. Point-of-Care Hemostatic Testing in Cardiac Surgery: A Stepped-Wedge Clustered Randomized Controlled Trial. Circulation. 2016 Oct 18;134(16):1152-1162. doi: 10.1161/CIRCULATIONAHA.116.023956. Epub 2016 Sep 21. PMID 27654344
- [Background] Kaufman RM, Djulbegovic B, Gernsheimer T, Kleinman S, Tinmouth AT, Capocelli KE, Cipolle MD, Cohn CS, Fung MK, Grossman BJ, Mintz PD, O'Malley BA, Sesok-Pizzini DA, Shander A, Stack GE, Webert KE, Weinstein R, Welch BG, Whitman GJ, Wong EC, Tobian AA; AABB. Platelet transfusion: a clinical practice guideline from the AABB. Ann Intern Med. 2015 Feb 3;162(3):205-13. doi: 10.7326/M14-1589. PMID 25383671
- [Background] Koch CG, Li L, Duncan AI, Mihaljevic T, Loop FD, Starr NJ, Blackstone EH. Transfusion in coronary artery bypass grafting is associated with reduced long-term survival. Ann Thorac Surg. 2006 May;81(5):1650-7. doi: 10.1016/j.athoracsur.2005.12.037. PMID 16631651
- [Background] Kwapisz MM, Kent B, DiQuinzio C, LeGare JF, Garnett S, Swyer W, Whynot S, Mingo H, Scheffler M. The prophylactic use of fibrinogen concentrate in high-risk cardiac surgery. Acta Anaesthesiol Scand. 2020 May;64(5):602-612. doi: 10.1111/aas.13540. Epub 2020 Jan 17. PMID 31889306
- [Background] Maquelin KN, Berckmans RJ, Nieuwland R, Schaap MC, ten Have K, Eijsman L, Sturk A. Disappearance of glycoprotein Ib from the platelet surface in pericardial blood during cardiopulmonary bypass. J Thorac Cardiovasc Surg. 1998 May;115(5):1160-5. doi: 10.1016/s0022-5223(98)70416-7. PMID 9605086
- [Background] Transfusion of Red Blood Cells, Fresh Frozen Plasma, or Platelets Is Associated With Mortality and Infection After Cardiac Surgery in a Dose-Dependent Manner. Anesth Analg. 2020 Feb;130(2):e32. doi: 10.1213/ANE.0000000000004528. PMID 31702696
- [Background] Ranucci M, Baryshnikova E, Castelvecchio S, Pelissero G; Surgical and Clinical Outcome Research (SCORE) Group. Major bleeding, transfusions, and anemia: the deadly triad of cardiac surgery. Ann Thorac Surg. 2013 Aug;96(2):478-85. doi: 10.1016/j.athoracsur.2013.03.015. Epub 2013 May 11. PMID 23673069
- [Background] Raphael J, Mazer CD, Subramani S, Schroeder A, Abdalla M, Ferreira R, Roman PE, Patel N, Welsby I, Greilich PE, Harvey R, Ranucci M, Heller LB, Boer C, Wilkey A, Hill SE, Nuttall GA, Palvadi RR, Patel PA, Wilkey B, Gaitan B, Hill SS, Kwak J, Klick J, Bollen BA, Shore-Lesserson L, Abernathy J, Schwann N, Lau WT. Society of Cardiovascular Anesthesiologists Clinical Practice Improvement Advisory for Management of Perioperative Bleeding and Hemostasis in Cardiac Surgery Patients. Anesth Analg. 2019 Nov;129(5):1209-1221. doi: 10.1213/ANE.0000000000004355. PMID 31613811
- [Background] Stanzel RD, Henderson M. Clinical evaluation of contemporary oxygenators. Perfusion. 2016 Jan;31(1):15-25. doi: 10.1177/0267659115604709. Epub 2015 Sep 25. PMID 26407816
- [Background] Weerasinghe A, Taylor KM. The platelet in cardiopulmonary bypass. Ann Thorac Surg. 1998 Dec;66(6):2145-52. doi: 10.1016/s0003-4975(98)00749-8. PMID 9930521